CLINICAL TRIAL: NCT01378208
Title: VEK-H-3-2011-023. Fasting and Meal Frequency Project
Brief Title: How Often Should We Eat
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Inge Holm (Other)
Responsible Party: Sponsor-Investigator, Inge Holm, CIM Administrator, Rigshospitalet, Denmark
Organization: Rigshospitalet, Denmark (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: VEK-H-3-2011-023
Record Dates: First submitted 2011-06-15; First posted 2011-06-22 (Estimated); Last update posted 2013-11-20 (Estimated); Status verified 2013-11

CONDITIONS: Intermittent Fasting; Meal Frequency
Keywords: Intermittent fasting; Meal frequency; body composition; cognitive function; glucose metabolism
MeSH Terms: conditions — Intermittent Fasting | interventions — Body Composition

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Normal weight (Experimental): Body Mass Index between 18-25 kg/m2 Age between 18-35 years male
  Interventions: Behavioral: Intermittent fasting - the effect on glucose metabolism, body composition and cognitive function

INTERVENTIONS:
Behavioral: Intermittent fasting - the effect on glucose metabolism, body composition and cognitive function — Each of the 10 subjects must through a period of monitoring (four weeks) before the study period (four weeks). Before, during, and after both the monitoring period and the study period, the subjects will undergo tests at Rigshospitalet.
  DAY 1: Inclusion and exclusion of subjects DAY 1 to DAY 28: Monitoring period (usual lifestyle)
  * 28 days of dietary monitoring
  * 28 days measurement by pedometer DAY 1, DAY 28 & DAY 56: Test 1
  * Oral glucose tolerance test with stable isotopes
  * Fat and muscle biopsies DAY 2, DAY 29 & DAY 57: Test 2
  * DXA scanning
  * Resting Metabolic Rate Measurement
  * VO2max test on bicycle
  * Cognitive testing
  * MRI of the brain and abdomen DAY 9, DAY 19, DAY 38 & DAY 48: Test 3
  * Actiheart for 3 days
  * 72-hour blood glucose monitoring with CGMS System DAY 29 to DAY 57: INTERVENTION
  * Fasting from 7am - 9pm
  * 28 days of dietary monitoring
  * 28 days measurement by pedometer

SUMMARY:
The Danish Food Administration recommends eating three main meals and three small meals a day in order to maintain a healthy lifestyle. However, there is little research to support this concept- moreover, many studies shows that fasting can have a positive impact on our health.

HYPOTHESIS AND PURPOSE The investigators hypothesize, that the number of meals per day in order to maintain a healthy lifestyle will not differ in normal weight subjects.

The investigators will include 1) healthy, normal weight subjects. The investigators will study the effects of two daily meals.

More specifically, the investigators want to better understand how the body reacts to long-term, intermittent fasting (14 h /day for 4 weeks). The investigators will assess cognitive function, dietary intake, appetite regulation, fitness, glucose and insulin responses, as well as fat and muscle composition of the body before, during, and after the study.

Our long-term goals are to compare the effects of intermittent fasting with acute fasting. All of this is in an effort to establish how our eating habits ultimately affect our health and to, perhaps, contribute to new recommendations for healthy eating in normal weight population.

BACKGROUND Obesity and diabetes are increasing health threats facing the Western world today, despite abundant research efforts and campaigns to prevent such outcomes. Throughout the years, as the incidence of both obesity and diabetes in the general population has increased, so too has the typical number of daily meals. A once common three meals per day has now increased to six meals per day, in many instances. Recent animal research has shown that intermittent fasting (one or two meals per day) over a long period of time can improve cardiovascular health and prevent chronic diseases. Biochemically, fasting leads to an activation of metabolic mechanisms designed to preserve carbohydrates and increase the dependence on energy produced by the metabolism of fat. There is little scientific evidence regarding the number of meals per day that proves to be the healthiest, and those studies that do exist have opposing conclusions. Several theories do exist regarding the number of meals per day that affect us in the most favorable way, but these are just theories. Our study is the first to assess, in both a systematic and controlled setting, how long-term, intermittent fasting affects the human body.

ELIGIBILITY:
Inclusion Criteria:

* Physically active, defined as at least 8,000 steps per day
* Regular meal frequency, i.e. energy intake=energy utilized, and eating between 3-6 meals per day

Exclusion Criteria:

* Daily medications
* Acute illness within the past two weeks (infection, fever, or surgery)
* Chronic disease, including cancer, heart, liver, kidney, and respiratory diseases, as well as metabolic diseases, such as diabetes
* Alcohol abuse or more than 14/21 units (women/men) consumed per week
* Smoking, including occasional smoking

Ages: 18 Years to 35 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 10 (Actual)
Dates: Start 2011-06; Primary Completion 2013-06 (Actual); Study Completion 2013-06 (Actual)

PRIMARY OUTCOMES:
oral glucose tolerance test and cognitive function | 2 months
  OGTT with stable isotopes. To see the effect of plasma glucose mmol/L and plasma insulin pmol/L 1 month after intervention (2 months from beginning of the study).
  Before, during, and after the intervention the subjects will complete cognitive tests for e.g. concentration, mood and appetite.

SECONDARY OUTCOMES:
Continuous glucose monitoring (CGM), body composition, and physical activity. | 2 months
  During the control period and the intervention the CGM system will measure the continuous glucose concentration (each 5 min), and thereby any change will be measured. Before, during, and after the intervention the subjects body composition will be determined by weight, hip, waist, and with DXA and MRI scans. Furthermore, physical activity will be assessed by Actiheart and VO2 max tests.

CONTACTS AND LOCATIONS:
Overall Officials: Bente K Pedersen, Professor, Study Director — Rigshospitalet, Denmark
Locations (1):
- Centre of Inflammation and Metabolism, Rigshospitalet, Copenhagen OE, Copenhagen, Denmark